CLINICAL TRIAL: NCT00853372
Title: Phase 2 Open-Label, Multi-Center Study to Evaluate the Safety and Efficacy of Sunitinib Malate in Combination With AMG 386 as First Line or Second Line Therapy for Subjects With Metastatic Renal Cell Carcinoma
Brief Title: AMG 386 Phase 2 Open-Label Renal Cell Carcinoma (RCC) Study 1st Line or After Cytokine Failure in Combination With Sunitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080579
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-05

CONDITIONS: Advanced Renal Cell Carcinoma
MeSH Terms: interventions — Sunitinib; trebananib; Angiogenesis Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trebananib 10 mg/kg + Sunitinib (Experimental): Trebananib 10 mg/kg intravenously (IV) once weekly (QW) plus sunitinib 50 mg orally (PO) once daily (QD) 4 weeks on/2 weeks off
  Interventions: Drug: Sunitinib; Drug: Trebananib
- Trebananib 15 mg/kg + Sunitinib (Experimental): Trebananib 15 mg/kg IV QW plus sunitinib 50 mg PO QD 4 weeks on/2 weeks off
  Interventions: Drug: Sunitinib; Drug: Trebananib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib will be administered 50 mg QD and is considered to be the background therapy as it is licensed for treatment of reneal cell cancer (RCC) and will be administered to all participants.
  Other Names: SUTENT (oral multi-kinase inhibitor)
Drug: Trebananib — Administered until a participant develops disease progression, clinical progression, unacceptable toxicity, withdraws consent, or death.
  Other Names: AMG 386; Angiogenesis inhibitor

SUMMARY:
This phase 2 study is an open-label, multi-center study to determine the safety and tolerability of AMG 386 in combination with sunitinib in the treatment of subjects with metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically confirmed metastatic renal cell cancer (RCC) with a clear cell component
* Low or intermediate risk according to the Memorial Sloan Kettering Cancer Center (MSKCC) prognostic risk classification
* Measurable disease with at least one unidimensionally measurable lesion per Response Evaluation Criteria in Solid Tumor (RECIST) guidelines with modifications
* Adequate organ and hematological function as evidenced by laboratory studies conducted at Screening
* Eastern Cooperative Oncology Group (ECOG) of 0 or 1

Exclusion Criteria:

Disease related

* Known history of central nervous system metastases.
* Previous treatment (excluding surgery, prior cytokine-based immunotherapy and palliative radiotherapy) for advanced or metastatic renal cell carcinoma
* Focal radiation therapy for palliation of pain from bony metastases within 14 days of enrollment.

Medications

* Currently or previously treated with sunitinib or other small molecule inhibitors of vascular endothelial growth factor (VEGF)
* Currently or previously treated with agents that neutralizing VEGF
* Currently or previously treated with AMG 386, or other molecules that inhibit the angiopoietins or Tie2 receptor
* Currently or previously treated with agents inhibiting the mammalian target of rapamycin (mTOR)
* Current or within 30 days prior to enrollment treatment with immune modulators
* Concomitant or previous use within 30 days prior to enrollment of any strong inducer of CYP3A4
* Concomitant or previous use of amiodarone within 6 months prior to enrollment

General medical

* Clinically significant cardiovascular disease within 12 months prior to enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication, percutaneous transluminal coronary angioplasty/stent
* Major surgery within 28 days prior to enrollment or still recovering from prior surgery
* Uncontrolled hypertension as defined as diastolic > 90 mmHg OR systolic >150 mmHg. The use of anti-hypertensive medications to control hypertension is permitted.

Other

* Other investigational procedures are excluded
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or subject is receiving other investigational agent(s)

Other inclusion/exclusion criteria may apply, per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-05-28 (Actual); Primary Completion 2011-08-08 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Atkins MB, Gravis G, Drosik K, Demkow T, Tomczak P, Wong SS, Michaelson MD, Choueiri TK, Wu B, Navale L, Warner D, Ravaud A. Trebananib (AMG 386) in Combination With Sunitinib in Patients With Metastatic Renal Cell Cancer: An Open-Label, Multicenter, Phase II Study. J Clin Oncol. 2015 Oct 20;33(30):3431-8. doi: 10.1200/JCO.2014.60.6012. Epub 2015 Aug 24. PMID 26304872
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 18 sites in the United States, Australia, Belgium, France, and Poland. The first participant was enrolled on 28 May 2009. The last participant was enrolled on 29 November 2010.
Period: Overall Study
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Started | 43 | 42
Completed | 11 | 13
Not Completed | 32 | 29
Not completed — Death | 30 | 26
Not completed — Lost to Follow-up | 1 | 2
Not completed — Full Consent Withdrawn | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Trebananib 10 mg/kg + Sunitinib: Trebananib 10 mg/kg IV QW plus sunitinib 50 mg PO QD 4 weeks on/2 weeks off
- Total: Total of all reporting groups
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Customized [Number; unit: participants]
  < 65 years | 30 | 27 | 57
  >= 65 years | 13 | 15 | 28
  < 75 years | 41 | 40 | 81
  >= 75 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 38 | 32 | 70
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 41 | 42 | 83
  Black or African American | 1 | 0 | 1
  Hispanic or Latino | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Japanese | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Aborigine | 0 | 0 | 0
  Other, Not Specified | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Discontinuations (DCs) Due to Adverse Events (AEs)
Description: AE: any untoward medical occurrence that does not necessarily have a causal relationship with treatment. SAE: an AE that: is fatal; is life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is an other significant medical hazard. Treatment-emergent AEs (TEAEs) are those that occurred after the first administration of study drug through 30 days after the last study drug administration. Severity was graded according to Common Terminology Criteria (CTCAE) version 3.0, as grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), grade 5 (death).
Time Frame: From first dose of study drug to 30 days after last dose. Median treatment duration of trebananib and sunitinib was 316 and 315 days, respectively, for Trebananib 10 mg/kg+Sunitinib, and 393 and 358 days, respectively, for Trebananib 15 mg/kg+Sunitinib.
Population: Safety Analysis Set: all participants who received at least 1 dose of trebananib and 1 dose of sunitinib.
Measure: Number; unit: participants
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 43 | 42
participants
  TEAEs, All | 43 | 42
  TEAEs, Grade ≥ 3 | 32 | 34
  TEAEs, Grade ≥ 4 | 4 | 7
  TEAEs, Fatal AEs | 1 | 1
  TEAEs, SAEs | 17 | 26
  TEAEs Leading to (→) DC of Trebananib | 7 | 14
  TEAEs → DC of Trebananib, Serious | 5 | 12
  TEAEs → DC of Trebananib, Non-Serious | 2 | 2
  TEAEs → DC of Sunitinib | 9 | 16
  TEAEs → DC of Sunitinib, Serious | 5 | 12
  TEAEs → DC of Sunitinib, Non-Serious | 4 | 5
  TEAEs → DC of All Treatment | 6 | 14
  TEAEs → DC of All Treatment, Serious | 5 | 12
  TEAEs → DC of All Treatment, Non-Serious | 1 | 2
  Treatment-Related (TR) TEAEs, All | 43 | 42
  TR TEAEs, Grade ≥ 3 | 25 | 31
  TR TEAEs, Grade ≥ 4 | 2 | 5
  TR TEAEs, Fatal AEs | 0 | 1
  TR TEAEs, SAEs | 11 | 18
  TR TEAEs → DC of Trebananib | 6 | 13
  TR TEAEs → DC of Trebananib, Serious | 4 | 11
  TR TEAEs → DC of Trebananib, Non-Serious | 2 | 2
  TR TEAEs → DC of Sunitinib | 8 | 15
  TR TEAEs → DC of Sunitinib, Serious | 4 | 11
  TR TEAEs → DC of Sunitinib, Non-Serious | 4 | 5
  TR TEAEs → DC of All Treatment | 5 | 13
  TR TEAEs → DC of All Treatment, Serious | 4 | 11
  TR TEAEs → DC of All Treatment, Non-Serious | 1 | 2
  Trebananib-Related (TrR) TEAEs, All | 34 | 39
  TrR TEAEs, Grade ≥ 3 | 17 | 19
  TrR TEAEs, Grade ≥ 4 | 1 | 4
  TrR TEAEs, Fatal AEs | 0 | 1
  TrR TEAEs, SAEs | 10 | 15
  TrR TEAEs → DC of Trebananib | 6 | 13
  TrR TEAEs → DC of Trebananib, Serious | 4 | 11
  TrR TEAEs → DC of Trebananib, Non-Serious | 2 | 2
  TrR TEAEs → DC of Sunitinib | 6 | 13
  TrR TEAEs → DC of Sunitinib, Serious | 4 | 11
  TrR TEAEs → DC of Sunitinib, Non-Serious | 2 | 3
  TrR TEAEs → DC of All Treatment | 5 | 13
  TrR TEAEs → DC of All Treatment, Serious | 4 | 11
  TrR TEAEs → DC of All Treatment, Non-Serious | 1 | 2
  Sunitinib-Related (SR) TEAEs, All | 43 | 42
  SR TEAEs, Grade ≥ 3 | 25 | 31
  SR TEAEs, Grade ≥ 4 | 2 | 5
  SR TEAEs, Fatal AEs | 0 | 1
  SR TEAEs, SAEs | 9 | 15
  SR TEAEs → DC of Trebananib | 4 | 11
  SR TEAEs → DC of Trebananib, Serious | 3 | 10
  SR TEAEs → DC of Trebananib, Non-Serious | 1 | 1
  SR TEAEs → DC Sunitinib | 7 | 13
  SR TEAEs → DC of Sunitinib, Serious | 3 | 10
  SR TEAEs → DC of Sunitinib, Non-Serious | 4 | 4
  SR TEAEs → DC of All Treatment | 4 | 11
  SR TEAEs → DC of All Treatment, Serious | 3 | 10
  SR TEAEs → DC of All Treatment, Non-Serious | 1 | 1

2. Primary Outcome: Number of Participants With Dose Delays Due to Adverse Events
Description: A trebananib dose was considered delayed if it was administered 11 or more days from the previous trebananib infusion. A sunitinib dose was considered delayed if it was administered 3 or more days from the previous dose, except during holidays.
Time Frame: Median treatment duration of trebananib and sunitinib was 316 and 315 days, respectively, for Trebananib 10 mg/kg+Sunitinib, and 393 and 358 days, respectively, for Trebananib 15 mg/kg+Sunitinib.
Population: Safety Analysis Set: participants who received at least 1 dose of trebananib and 1 dose of sunitinib.
Measure: Number; unit: participants
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 43 | 42
participants
  Trebananib Dose Delays | 26 | 28
  Sunitinib Dose Delays | 29 | 27

3. Primary Outcome: Number of Participants With Sunitinib Dose Modifications Within 12 Weeks of First Dose
Description: Participants who had a sunitinib dose modification within 12 weeks from their first dose due to adverse event, laboratory toxicity, or laboratory toxicity and adverse event.
Time Frame: first 12 weeks of study treatment
Population: Safety Analysis Set: all participants who received at least 1 dose of trebananib and 1 dose of sunitinib.
Measure: Number; unit: participants
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 43 | 42
participants
  Any Dose Modification (DM) | 25 | 24
  DM Due to Adverse Event | 20 | 18
  DM Due to Laboratory Toxicity | 4 | 4
  DM Due to Laboratory Toxicity and Adverse Event | 1 | 2

4. Primary Outcome: Number of Participants With Worst Post-Baseline Grade 3 or Higher Toxicity in Laboratory Values
Description: Severity was graded according to Common Terminology Criteria (CTCAE) version 3.0, as grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), grade 5 (death).
Time Frame: as for outcome 1
Population: Safety Aanalysis Set: all participants who received at least 1 dose of trebananib and 1 dose of sunitinib.
Measure: Number; unit: participants
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 43 | 42
participants
  Alanine Aminotransferase, Above Normal (AN) | 3 | 2
  Albumin, Below Normal (BN) | 1 | 1
  Alkaline Phosphatase, AN | 0 | 2
  Amylase, AN | 2 | 5
  Aspartate Aminotransferase, AN | 2 | 2
  Glucose, AN | 1 | 3
  Glucose, BN | 1 | 0
  Lipase, AN | 5 | 7
  Magnesium, BN | 0 | 1
  Phosphorus, BN | 3 | 4
  Potassium, BN | 2 | 2
  Sodium, BN | 1 | 4
  Total Bilirubin, AN | 0 | 2
  Absolute Neutrophil Count, BN | 3 | 5
  Hemoglobin, BN | 1 | 3
  Lymphocytes, BN | 6 | 3
  Partial Thromboplastin Time, AN | 1 | 1
  Platelets, BN | 3 | 2
  Total Neutrophils, BN | 3 | 5

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with either a confirmed complete response (CR) or partial response (PR) per modified Response Evaluation Criteria in Solid Tumor (RECIST) criteria (responder). A confirmed CR requires 2 consecutive assessments of CR at least 28 days apart. A confirmed PR requires 2 consecutive assessments at least 28 days apart of PR or CR. All participants who did not meet the criteria for an objective response by the analysis cutoff date were considered non responders.
Time Frame: 48 months after last subject enrolled (LSE)
Population: Safety Analysis Set: all participants who received at least 1 dose of trebananib and 1 dose of sunitinib. Participants with baseline measureable disease.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 43 | 41
percentage of participants | 58.1 [47.2 to 68.5] | 63.4 [52.2 to 73.6]

6. Secondary Outcome: Kaplan-Meier Estimate: Duration of Response (DOR)
Description: DOR was calculated as the time from the first confirmed objective response to first observed disease progression per modified RECIST v. 1.0 criteria or death due to any cause. DOR was calculated only for participants who had an objective response. Objective response was defined as either a confirmed CR or PR per modified RECIST criteria. A confirmed CR required 2 consecutive assessments of CR at least 28 days apart. A confirmed PR required 2 consecutive assessments at least 28 days apart of PR or CR.
  Participants not meeting criteria for progression by the analysis data cutoff date were censored at their last evaluable radiographical disease assessment date.
Time Frame: 48 months after LSE
Population: Safety Analysis Set: all participants who received at least 1 dose of trebananib and 1 dose of sunitinib. Participants with an objective response.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 25 | 26
months | 18.0 [11.8 to 24.4] | 18.4 [11.5 to 24.8]

7. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with confirmed CR or PR or stable disease (SD), as defined by modified RECIST v1.0 criteria. A confirmed CR required 2 consecutive assessments of CR at least 28 days apart. A confirmed PR requires 2 consecutive assessments at least 28 days apart of PR or CR. CR or PR was confirmed at least 28 days after the criteria for response were first met. A response assessment of PR or CR that was not subsequently confirmed at least 4 weeks later were included as SD.
Time Frame: 48 months after LSE
Population: as for outcome 5
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 43 | 41
percentage of participants | 72.1 [61.5 to 81.0] | 75.6 [64.9 to 84.3]

8. Secondary Outcome: Kaplan-Meier Estimate: Progression Free Survival (PFS)
Description: PFS was defined as the time from enrollment date to date of disease progression (ie, radiographic progression) per modified RECIST v 1.0 criteria or death. Radiological imaging to assess disease status was performed until participants developed disease progression. Events of radiographic progression per modified RECIST 1.0 that occurred after initiation of subsequent anticancer therapy were not considered PFS events. Deaths occurring after initiation of subsequent anticancer therapy were considered PFS events.
  Participants not meeting criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Time Frame: 48 months after LSE
Population: Safety Analysis Set: all participants who received at least 1 dose of trebananib and 1 dose of sunitinib.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 43 | 42
months | 13.9 [11.0 to 16.1] | 16.5 [13.3 to 21.4]

9. Secondary Outcome: Kaplan-Meier Estimate: Overall Survival (OS)
Description: The time from enrollment date to date of death. Participants who had not died by the analysis data cutoff date were censored at their last contact date.
Time Frame: 48 months after LSE
Population: Safety Analysis Set: all participants who received at least 1 dose of trebananib and 1 dose of sunitinib.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 43 | 42
months | 36.0 [26.0 to 52.9] | 38.7 [31.5 to 42.6]

10. Secondary Outcome: Maximum Percent Reduction From Baseline in the Sum of the Longest Diameters (SLD) of Target Lesions From Baseline to Post-Baseline Nadir
Description: Change in tumor burden was evaluated by the maximum percent reduction from baseline in the SLD of target lesions.
Time Frame: Baseline, 48 months after LSE
Population: Safety Analysis Set: all participants who received at least 1 dose of trebananib and 1 dose of sunitinib. Participants with baseline measureable disease and non-missing baseline and post-baseline data.
Measure: Mean (80% Confidence Interval); unit: percent reduction in SLD
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 41 | 40
percent reduction in SLD | -36.0 [-43.4 to -28.6] | -41.8 [-48.4 to -35.3]

11. Secondary Outcome: Pharmacokinetic Parameter: Maximum Observed Concentration (Cmax) for Trebananib Over Time
Time Frame: Pre-infusion and up to 10 minutes post-infusion on Weeks 1, 4, 7, 10, 13, 22, 34, 46, 58, 70, 82, 94, 106, and safety follow-up (30 ±7 days after the last dose of study drug)
Population: Pharmacokinetics Analysis Set: participants with evaluable concentration data at given time point.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 38 | 41
µg/mL
  Week 1 | 222 [63.2 to 819] | 297 [152 to 535]
  Week 4: number analyzed (Participants) | 32 | 22
  Week 4 | 285 [82.4 to 574] | 377 [258 to 647]
  Week 7: number analyzed (Participants) | 32 | 28
  Week 7 | 260 [75.3 to 550] | 377 [238 to 1830]
  Week 10: number analyzed (Participants) | 32 | 23
  Week 10 | 257 [105 to 630] | 476 [184 to 770]
  Week 13: number analyzed (Participants) | 26 | 22
  Week 13 | 219 [105 to 390] | 385 [216 to 785]
  Week 22: number analyzed (Participants) | 31 | 23
  Week 22 | 249 [92.8 to 385] | 417 [224 to 758]
  Week 34: number analyzed (Participants) | 24 | 18
  Week 34 | 240 [137 to 628] | 387 [77.7 to 571]
  Week 46: number analyzed (Participants) | 19 | 7
  Week 46 | 221 [159 to 700] | 349 [235 to 908]
  Week 58: number analyzed (Participants) | 13 | 0
  Week 58 | 229 [158 to 606] |
  Week 70: number analyzed (Participants) | 15 | 0
  Week 70 | 185 [108 to 362] |
  Week 82: number analyzed (Participants) | 6 | 0
  Week 82 | 223 [94.1 to 272] |
  Week 94: number analyzed (Participants) | 2 | 0
  Week 94 | 270 [173 to 367] |
  Week 106: number analyzed (Participants) | 1 | 0
  Week 106 | 289 [289 to 289] |
  Safety Follow-Up: number analyzed (Participants) | 11 | 3
  Safety Follow-Up | 3.46 [1.26 to 6.16] | 8.26 [5.62 to 11.8]

12. Secondary Outcome: Pharmacokinetic Parameter: Minimum Observed Concentration (Cmin) for Trebananib Over Time
Time Frame: Pre-infusion on Weeks 4, 7, 10, 13, 22, 34, 46, 58, 70, 82, 94, 106, and safety follow-up (30 ±7 days after the last dose of study drug)
Population: Pharmacokinetics Analysis Set: participants with evaluable concentration data at given time point.
Measure: Median (Full Range); unit: µg/mL
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 38 | 29
µg/mL
  Week 4 | 20.4 [6.22 to 41.9] | 27.3 [6.35 to 95.4]
  Week 7: number analyzed (Participants) | 35 | 29
  Week 7 | 30.1 [12.2 to 75.9] | 42.0 [14.9 to 90.4]
  Week 10: number analyzed (Participants) | 33 | 23
  Week 10 | 23.3 [9.09 to 72.3] | 32.2 [13.9 to 85.6]
  Week 13: number analyzed (Participants) | 33 | 25
  Week 13 | 26.1 [8.54 to 73.8] | 43.2 [15.1 to 99.5]
  Week 22: number analyzed (Participants) | 32 | 24
  Week 22 | 19.9 [8.59 to 63.1] | 46.2 [16.2 to 73.7]
  Week 34: number analyzed (Participants) | 23 | 18
  Week 34 | 24.1 [9.88 to 66.2] | 35.9 [15.3 to 79.2]
  Week 46: number analyzed (Participants) | 21 | 8
  Week 46 | 23.2 [6.46 to 64.4] | 30.5 [21.0 to 71.8]
  Week 58: number analyzed (Participants) | 15 | 0
  Week 58 | 27.9 [8.61 to 43.3] |
  Week 70: number analyzed (Participants) | 15 | 0
  Week 70 | 26.2 [10.5 to 35.9] |
  Week 82: number analyzed (Participants) | 5 | 0
  Week 82 | 22.5 [17.9 to 33.0] |
  Week 94: number analyzed (Participants) | 2 | 0
  Week 94 | 25.9 [19.9 to 31.8] |
  Week 106: number analyzed (Participants) | 1 | 0
  Week 106 | 19.3 [19.3 to 19.3] |
  Safety Follow-Up: number analyzed (Participants) | 11 | 3
  Safety Follow-Up | 3.46 [1.26 to 6.16] | 8.26 [5.62 to 11.8]

13. Secondary Outcome: Pharmacokinetic Parameter: Cmin for Sunitinib Over Time
Time Frame: Pre-infusion on Weeks 4, 7, 10, 16, 22, 34, 46, 58, 70, 82, 94, 106, and safety follow-up (30 ±7 days after the last dose of study drug)
Population: Pharmacokinetics Analysis Set: participants with evaluable concentration data at given time point. Per protocol, this outcome measure evaluated a sub-group of participants at selected sites outside of Europe.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 9 | 7
ng/mL
  Week 4: number analyzed (Participants) | 6 | 6
  Week 4 | 58.6 [41.1 to 124] | 70.6 [50.8 to 105]
  Week 7 | 0.763 [NA to 4.68] — below lower limit of quantification (0.25 ng/mL) | 1.65 [NA to 3.78] — below lower limit of quantification (0.25 ng/mL)
  Week 10: number analyzed (Participants) | 9 | 5
  Week 10 | 66.1 [46.7 to 136] | 64.7 [42.4 to 95.4]
  Week 16: number analyzed (Participants) | 5 | 3
  Week 16 | 65.8 [47.1 to 91.9] | 73.1 [49.1 to 92.7]
  Week 22: number analyzed (Participants) | 5 | 1
  Week 22 | 49.0 [33.3 to 97.1] | 41.2 [41.2 to 41.2]
  Week 34: number analyzed (Participants) | 4 | 1
  Week 34 | 50.2 [NA to 110] — below lower limit of quantification (0.25 ng/mL) | 34.8 [34.8 to 34.8]
  Week 46: number analyzed (Participants) | 3 | 2
  Week 46 | 59.5 [49.4 to 66.4] | 33.5 [23.3 to 43.7]
  Week 58: number analyzed (Participants) | 2 | 0
  Week 58 | 87.0 [51.9 to 122] |
  Week 70: number analyzed (Participants) | 1 | 0
  Week 70 | 56.4 [56.4 to 56.4] |
  Week 82: number analyzed (Participants) | 1 | 0
  Week 82 | 65.9 [65.9 to 65.9] |
  Week 94: number analyzed (Participants) | 1 | 0
  Week 94 | 64.2 [64.2 to 64.2] |
  Week 106: number analyzed (Participants) | 1 | 0
  Week 106 | 83.5 [83.5 to 83.5] |
  Safety Follow-Up: number analyzed (Participants) | 6 | 0
  Safety Follow-Up | NA [NA to 2.14] — below lower limit of quantification (0.25 ng/mL) |

14. Secondary Outcome: Pharmacokinetic Parameter: Cmin for Sunitinib Metabolite Over Time
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 9 | 7
ng/mL
  Week 4: number analyzed (Participants) | 6 | 6
  Week 4 | 22.8 [11.6 to 29.4] | 29.2 [16.5 to 43.4]
  Week 7 | 1.21 [0.582 to 3.89] | 1.71 [0.405 to 3.22]
  Week 10: number analyzed (Participants) | 9 | 5
  Week 10 | 19.2 [14.0 to 40.6] | 21.5 [18.0 to 41.3]
  Week 16: number analyzed (Participants) | 5 | 3
  Week 16 | 19.3 [13.7 to 22.7] | 22.0 [21.6 to 40.5]
  Week 22: number analyzed (Participants) | 5 | 1
  Week 22 | 12.7 [10.1 to 28.5] | 18.7 [18.7 to 18.7]
  Week 34: number analyzed (Participants) | 4 | 1
  Week 34 | 18.3 [NA to 38.3] — below lower limit of quantification (0.25 ng/mL) | 15.0 [15.0 to 15.0]
  Week 46: number analyzed (Participants) | 3 | 2
  Week 46 | 15.0 [10.3 to 23.1] | 10.6 [7.87 to 13.4]
  Week 58: number analyzed (Participants) | 2 | 0
  Week 58 | 25.7 [20.1 to 31.2] |
  Week 70: number analyzed (Participants) | 1 | 0
  Week 70 | 22.4 [22.4 to 22.4] |
  Week 82: number analyzed (Participants) | 1 | 0
  Week 82 | 25.4 [25.4 to 25.4] |
  Week 94: number analyzed (Participants) | 1 | 0
  Week 94 | 22.1 [22.1 to 22.1] |
  Week 106: number analyzed (Participants) | 1 | 0
  Week 106 | 32.4 [32.4 to 32.4] |
  Safety Follow-Up: number analyzed (Participants) | 6 | 0
  Safety Follow-Up | 0.138 [NA to 1.15] — below lower limit of quantification (0.25 ng/mL) |

15. Secondary Outcome: Number of Participants Binding Antibody- or Neutralizing Antibody-Positive Post-Baseline
Description: Transient positive results were defined as a positive post-baseline result followed by a negative result at the participant's last time point tested within the study period.
Time Frame: 48 months after LSE
Population: Safety Analysis Set: all participants who received at least 1 dose of trebananib and 1 dose of sunitinib. Participants with a post-baseline result and a negative result or no result at baseline.
Measure: Number; unit: participants
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Number analyzed (Participants) | 41 | 41
participants
  Binding Antibody Positive Post-Baseline (PBL) | 0 | 0
  Binding Antibody Positive PBL, Transient | 0 | 0
  Neutralizing Antibody Positive PBL | 0 | 0
  Neutralizing Antibody Positive PBL, Transient | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after last dose. Median treatment duration of trebananib and sunitinib was 316 and 315 days, respectively, for Trebananib 10 mg/kg+Sunitinib, and 393 and 358 days, respectively, for Trebananib 15 mg/kg+Sunitinib.
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. Other adverse events shows non-serious occurrences of adverse event that exceed the indicated frequency threshold.
Arm/Group | Trebananib 10 mg/kg + Sunitinib | Trebananib 15 mg/kg + Sunitinib
Serious Adverse Events (participants affected / at risk) | 17/43 | 26/42
Other Adverse Events (participants affected / at risk) | 43/43 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trebananib 10 mg/kg + Sunitinib (N=43) | Trebananib 15 mg/kg + Sunitinib (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Papilloedema (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Rectourethral fistula (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 3
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 2 | 1
Infusion site inflammation (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Mucosal inflammation (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Swelling (General disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain hypoxia (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Migraine with aura (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Device occlusion (Product Issues) | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trebananib 10 mg/kg + Sunitinib (N=43) | Trebananib 15 mg/kg + Sunitinib (N=42)
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Leukopenia (Blood and lymphatic system disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 5 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 11
Pericardial effusion (Cardiac disorders) | 1 | 3
Hypoacusis (Ear and labyrinth disorders) | 3 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 4
Hyperthyroidism (Endocrine disorders) | 2 | 5
Hypothyroidism (Endocrine disorders) | 21 | 18
Eyelid oedema (Eye disorders) | 10 | 8
Glaucoma (Eye disorders) | 3 | 0
Lacrimation increased (Eye disorders) | 13 | 12
Periorbital oedema (Eye disorders) | 5 | 8
Visual acuity reduced (Eye disorders) | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 15
Abdominal pain upper (Gastrointestinal disorders) | 14 | 9
Aphthous ulcer (Gastrointestinal disorders) | 9 | 6
Ascites (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 13 | 8
Diarrhoea (Gastrointestinal disorders) | 33 | 32
Dry mouth (Gastrointestinal disorders) | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 16 | 10
Dysphagia (Gastrointestinal disorders) | 1 | 5
Flatulence (Gastrointestinal disorders) | 2 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 3
Gingival pain (Gastrointestinal disorders) | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 22 | 19
Oesophagitis (Gastrointestinal disorders) | 1 | 3
Stomatitis (Gastrointestinal disorders) | 4 | 8
Vomiting (Gastrointestinal disorders) | 17 | 13
Asthenia (General disorders) | 16 | 20
Catheter site pain (General disorders) | 3 | 0
Chest pain (General disorders) | 1 | 5
Chills (General disorders) | 3 | 6
Face oedema (General disorders) | 15 | 21
Fatigue (General disorders) | 16 | 14
Generalised oedema (General disorders) | 4 | 3
Influenza like illness (General disorders) | 2 | 3
Localised oedema (General disorders) | 6 | 3
Malaise (General disorders) | 4 | 1
Mucosal dryness (General disorders) | 3 | 0
Mucosal inflammation (General disorders) | 22 | 25
Oedema peripheral (General disorders) | 24 | 24
Pyrexia (General disorders) | 4 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 3
Bronchitis (Infections and infestations) | 3 | 3
Conjunctivitis (Infections and infestations) | 4 | 4
Cystitis (Infections and infestations) | 0 | 3
Ear infection (Infections and infestations) | 1 | 3
Gastroenteritis (Infections and infestations) | 6 | 1
Influenza (Infections and infestations) | 4 | 1
Laryngitis (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 4 | 2
Oral herpes (Infections and infestations) | 3 | 2
Pharyngitis (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 8 | 4
Sinusitis (Infections and infestations) | 2 | 3
Tooth abscess (Infections and infestations) | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 7
Urinary tract infection (Infections and infestations) | 1 | 4
Fall (Injury, poisoning and procedural complications) | 4 | 0
Alanine aminotransferase increased (Investigations) | 3 | 3
Amylase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 2
Blood creatinine increased (Investigations) | 3 | 3
Lipase increased (Investigations) | 1 | 5
Weight decreased (Investigations) | 5 | 4
Weight increased (Investigations) | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 17 | 24
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 8
Obesity (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 5
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Ageusia (Nervous system disorders) | 5 | 3
Dizziness (Nervous system disorders) | 10 | 6
Dysgeusia (Nervous system disorders) | 6 | 3
Formication (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 13 | 6
Neuropathy peripheral (Nervous system disorders) | 3 | 4
Paraesthesia (Nervous system disorders) | 3 | 3
Presyncope (Nervous system disorders) | 4 | 1
Sciatica (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 1 | 3
Taste disorder (Nervous system disorders) | 14 | 10
Anxiety (Psychiatric disorders) | 4 | 2
Depression (Psychiatric disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 8 | 5
Dysuria (Renal and urinary disorders) | 3 | 5
Proteinuria (Renal and urinary disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 6
Erythema (Skin and subcutaneous tissue disorders) | 6 | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 5 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 21 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 9 | 9
Skin discolouration (Skin and subcutaneous tissue disorders) | 4 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 3 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 | 3
Skin toxicity (Skin and subcutaneous tissue disorders) | 4 | 4
Yellow skin (Skin and subcutaneous tissue disorders) | 4 | 5
Hypertension (Vascular disorders) | 26 | 23
Hypotension (Vascular disorders) | 3 | 7
Pallor (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.